CLINICAL TRIAL: NCT00743054
Title: microRNA Expression in Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: SYSU-MiRNARCC
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Carcinoma, Renal Cell
Keywords: Carcinoma, Renal Cell; MicroRNAs
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The tumor tissues and tumor adjacent tissues will be collected when patients receive renal cell carcinoma resection.
  The blood and urine will be collected before patients receive operation. And the blood and urine of some healthy volunteers will be collected as the control group.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, renal cell carcinoma (RCC) related miRNA and the target genes of related miRNA will be examined in order to investigate the role of miRNA in the formation of RCC and look for the biomarker of RCC.

DETAILED DESCRIPTION:
Due to the lack of specific indicators for the early diagnosis of RCC, the RCC patients often have distant metastasis when diagnosed and their five-year survival rate is much low. Therefore, the biological markers of RCC are needed for early detection, early treatment and improvement of the survival rate of RCC patients.

MiRNA and tumor are closely related. MiRNA can control the important cancer-related genes and participate in the tumor cell proliferation, apoptosis, invasion and angiogenesis.

In this study, RCC related miRNA and the target genes of related miRNA will be examined,and the relationship between RCC related miRNA and the RCC pathological types, TNM (tumor-nodes-metastasis) stages and prognosis will be analyzed. The purpose of this study is to investigate the role of miRNA in the formation of RCC and look for the biomarker of RCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary renal cell carcinoma.
* Subjects who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients with secondary renal cell carcinoma.
* Subjects who refuse to participate in the study and sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients in the department of Urology of 1st Affiliated Hospital, Sun Yat-Sen University
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China